CLINICAL TRIAL: NCT06840600
Title: Public Support for Prison Nutrition Standards
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 25-0030
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-05

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Public safety rationale (Experimental)
  Interventions: Behavioral: Public safety rationale
- Right-to-health rationale (Experimental)
  Interventions: Behavioral: Right-to-health rationale
- Cost-saving rationale (Experimental)
  Interventions: Behavioral: Cost-saving rationale
- No rationale (Control) (Other)
  Interventions: Behavioral: No rationale (Control)

INTERVENTIONS:
Behavioral: Public safety rationale — Rationale provided for policy is to increase community safety.
  Arms: Public safety rationale
Behavioral: Right-to-health rationale — Rationale provided for policy is to support humans' right to healthy food.
  Arms: Right-to-health rationale
Behavioral: Cost-saving rationale — Rationale provided for policy is to save the government money.
  Arms: Cost-saving rationale
Behavioral: No rationale (Control) — In this arm, no rationale is provided for the policy.
  Arms: No rationale (Control)

SUMMARY:
The goal of this experiment is to examine the impact of policy rationale on public support for prison nutrition standards. The main question this experiment aims to answer is:

Does the rationale provided for a policy to improve prison nutrition standards impact public support for such a policy?

Additionally, this experiment aims to answer:

To what extent are participant demographic characteristics correlated with public support for prison nutrition standards?

DETAILED DESCRIPTION:
This study aims to examine the impact of policy rationale on public support for prison nutrition standards. In an online survey, participants will be asked to imagine a new U.S. policy which would require prisons to serve meals that meet the government definition of healthy. Participants will then be randomly assigned to view 1 of 3 different rationales for the new policy, or be assigned to a control arm where no rationale is given. All participants will answer a question about support for the policy.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Report residing in the US
* Can read and speak English
* Have internet access to complete the online survey

Exclusion Criteria:

* Under 18 years of age
* Residing outside the US

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1201 (Actual)
Dates: Start 2025-05-07 (Actual); Primary Completion 2025-06-04 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
Policy Support | Assessed one-time via online survey immediately after participant views each policy rationale (exposure to study stimuli). Overall survey will take approximately 15 minutes.
  Policy support will be measured with an item that reads "Would you…" with response options on a 5-point scale ranging from "Strongly oppose this law" coded as 1, to "Strongly support this law", coded as 5. Higher scores indicate stronger policy support.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Chelius, MS, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-03-26): https://cdn.clinicaltrials.gov/large-docs/00/NCT06840600/SAP_000.pdf